CLINICAL TRIAL: NCT01515709
Title: Is the Short Physical Performance Battery a Useful Outcome Measure in Patients With Chronic Obstructive Pulmonary Disease ?
Brief Title: Is the Short Physical Performance Battery a Useful Outcome Measure in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011LF001H
Record Dates: First submitted 2012-01-10; First posted 2012-01-24 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Pulmonary Emphysema; Bronchitis, Chronic; Lung Diseases; Disease Progression
Keywords: Cohort Studies; Longitudinal Studies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Pulmonary Emphysema; Bronchitis, Chronic; Lung Diseases; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: Patients with a diagnosis of COPD

SUMMARY:
Patients with Chronic Obstructive Lung Disease (COPD) often develop muscle problems, particularly in their legs which makes them more limited in what they can do. The Short Physical Performance Battery (SPPB) is a simple test of standing balance, usual walking speed and ability to stand from a chair. The SPPB may be a useful measure to predict leg function.

This study aims to evaluate whether the SPPB is comparable with current exercise tests used in COPD patients, and whether it is useful in predicting disability, death and health resource usage over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD

Exclusion Criteria:

* Any patient in whom mobility and lower limb function have been significantly affected by a neuromuscular cause (eg. motor neurone disease), severe peripheral vascular disease or amputation
* Any patient whom is deemed unsafe to exercise
* Patients unable to complete the SPPB, walking tests and leg strength assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a diagnosis of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 36 months

SECONDARY OUTCOMES:
Hospitalisation rate | 36 months
Healthcare resource usage | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MRCP PhD, Principal Investigator — NIHR Respiratory Biomedical Research Unit, Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Harefield, United Kingdom

REFERENCES:
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Derived] Nolan CM, Kon SSC, Patel S, Jones SE, Barker RE, Polkey MI, Maddocks M, Man WD. Gait speed and pedestrian crossings in COPD. Thorax. 2018 Feb;73(2):191-192. doi: 10.1136/thoraxjnl-2017-210173. Epub 2017 May 5. PMID 28476882